CLINICAL TRIAL: NCT06937242
Title: Fall-related Health Outcome in Lower Limb Prosthesis Users: A Pragmatic Clinical Trial to Assess Effectiveness of Microprocessor-controlled Prosthetic Knees
Brief Title: Effects of Microprocessor-controlled Prosthetic Knees on Fall-related Health Outcomes in Limited Community Ambulators
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanger Institute for Clinical Research and Education, LLC (Industry)
Collaborators: University of Washington (Other); U.S. Army Medical Research Acquisition Activity (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: UW-724; CDMRP-CDMRP Log OP190025 (Other Grant/Funding Number: US Department of Defense (DOD), Grant Office)
Record Dates: First submitted 2025-04-11; First posted 2025-04-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Amputation; Prosthesis User; Amputation; Traumatic, Leg: Thigh, Between Hip and Knee; Limb; Absence, Congenital, Lower; Lower Limb Amputation Above Knee (Injury); Lower Limb Amputation Above Knee
Keywords: amputation; lower limb amputation; lower limb prosthesis user; mechanical knee; microprocessor knee; transfemoral amputation; knee disarticulation; prosthetic knee; falls; falling; amputee; transfemoral amputee; MPK
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to the intervention or control group. Participants randomized to the intervention arm of the trial will have their nMPK exchanged for either a stance-and-swing MPK (Ottobock C-Leg 4) or a stance-only MPK (Ottobock Kenevo). Participants in the control arm of the trial will remain in their prescribed prosthesis with a nMPK.
Who Masked: Participant, Care Provider
Masking Description: The randomization plan will be hidden from investigators responsible for enrolling and consenting study participants. The prosthetist and participant will be unblinded to assignment following enrollment. It is not feasible to blind participants throughout the study due to key differences in the intervention and control devices (e.g., the MPK requires daily charging, but the NMPK does not).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MPK (Ottobock C-Leg 4 or Ottobock Kenevo) (Experimental): The MPK provided to each participant in the intervention arm will be determined by the manufacturer's recommended patient-selection criteria.
  Interventions: Device: Ottobock C-Leg 4 Microprocessor Knee; Device: Ottobock Kenevo
- nMPK (No Intervention): Participants in the control arm of the trial will remain in their prescribed non-microprocessor knee (nMPK) prosthesis

INTERVENTIONS:
Device: Ottobock C-Leg 4 Microprocessor Knee — Subjects in the intervention group who can walk more than 0.83m/s in the 2-minute walk test (2MWT) will receive the Ottobock C-Leg 4, a stance-and-swing microprocessor knee.
  Arms: MPK (Ottobock C-Leg 4 or Ottobock Kenevo)
Device: Ottobock Kenevo — Subjects in the intervention group who can walk up to 0.83m/s (3km/hr) in the 2-minute walk test (2MWT) will receive the Kenevo, a stance-only microprocessor knee.
  Arms: MPK (Ottobock C-Leg 4 or Ottobock Kenevo)

SUMMARY:
The goal of this study is to find out if using microprocessor-controlled prosthetic knees (MPKs), prosthetic knees with a built-in computer, improves health outcomes related to falls in adults who use above-knee prostheses. The main questions are:

* Do individuals with MPKs have fewer fall-related health issues compared to those with non-microprocessor-controlled prosthetic knees (nMPKs)?
* Do individuals with MPKs have increased mobility, faster walking speed, and improved quality of life compared to those with nMPKs?

Participants who have recently received an nMPK as part of their regular care can join the study. Those randomized to the control group will keep using their nMPK, while those randomized to the intervention group will receive a stance-and-swing MPK or a stance-only MPK.

DETAILED DESCRIPTION:
This study aims to assess the effects of microprocessor-controlled prosthetic knees on fall-related health outcomes in prosthesis users classified as limited community ambulators. This study also seeks to expand the existing research on the potential microprocessor-controlled prosthetic knees (MPKs) have on improving health outcomes for patients who are classified as limited community ambulators (i.e., Medicare Functional Level K2). The investigators will examine whether the anticipated reduction in falls in K2 users is accompanied by improvements in fall-related health outcomes like fall-related anxiety, fall-related self-efficacy, fall-related avoidance behaviors, fall-related interference, and fewer falls. Investigators will also examine whether MPK use in the K2 population leads to increased mobility, increased walking speed, and improvements in health-related quality of life.

A 12-month, pragmatic randomized control trial (pRCT) will be conducted to assess whether MPKs improve fall-related health outcomes in unilateral, transfemoral or knee disarticulation prosthesis users classified as limited community ambulators.

Patients will be invited to participate in the trial as a part of their routine prosthetic care. If a patient agrees to participate and is eligible, a follow-up appointment will be scheduled, and the patient will be consented by the research study team. Participants will then be randomized to the intervention or control group. Participants in the control arm of the trial will remain in their prescribed prosthesis with a non-microprocessor knee (nMPK). Participants randomized to the intervention arm of the trial will have their nMPK exchanged for either a stance-and-swing MPK (Ottobock C-Leg 4) or a stance-only MPK (Ottobock Kenevo). The MPK provided to each participant in the intervention arm will be determined by the manufacturer's recommended patient-selection criteria. Transfemoral prosthesis users walking up to 0.83m/s (3km/hr) in the 2-minute walk test (2MWT) will receive a stance-only MPK (Kenevo), while participants walking more than 0.83m/s in the 2MWT will receive a stance-and-swing MPK (C-Leg 4). Study participants will wear the knee for 12 months.

Each participant will be assessed at baseline (after enrollment and randomization), and 1-, 3-, 6-, 9-, and 12-months after baseline. The baseline and 12-month assessments will be the primary study time points. T-scores on the Prosthetic Limb Users Survey of Fall-Related Health (PLUS-F) and number of fall events experienced over the prior year will serve as the primary endpoints. Participants will complete a selected set of performance-based tests and standardized self-report surveys. In addition to the outcome measures noted, investigators will collect sociodemographic, health, amputation, fall history, and prosthesis information by self-report in order to characterize study participants and assess the comparability of the study groups. Fall-related health outcomes (e.g. fall-related self-efficacy and fall-related interference) will be measured using new PLUS-F instruments as well as existing measures that measure fall-related outcomes. We will also co-administer the Prosthetic Limb Users Survey of Mobility (PLUS-M) to assess participants' prosthesis-related mobility. Walking speed, mobility, endurance, and quality of life will be measured. For the 6- and 12-month assessments, we will also collect the hours of wear and hours of activity in the prosthesis.

Participants in both groups will receive education and training specific to their prosthetic knee between assessment 1 (baseline) and assessment 2 (one-month follow-up). Training will consist of 1 to 4 sessions to facilitate participants' use of their assigned prostheses. The number of sessions will be determined by the ability of each participant to explain and/or perform specified tasks. A standardized protocol and training checklist will be developed by our team Physical Therapist specific to each condition in collaboration with the knees' manufacturer (Ottobock). Every 2 weeks, throughout the 12 months of patient participation, the number of falls and near-fall events, including the event, injury, treatment and/or hospitalization, and whether the falls occurred while wearing the prosthesis, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transfemoral or knee disarticulation limb loss.
* 6 months or longer since time of limb loss.
* Current user of a prosthesis with a non-microprocessor-controlled prosthetic knee.
* Received a replacement prosthesis with a non-microprocessor knee in the past 4-24 months.
* Clinician has deemed patient limited community ambulator (Medicare functional classification level K2).
* In addition, Medicare functional classification level K2 as determined by at least one of the following criteria:

  1. Houghton Score: 5-10
  2. Prosthetic Limb Users Survey of Mobility (PLUS-M) T-Score: if amputation etiology is vascular disease/diabetes <49.45, otherwise, <36.75.
  3. Amputee Mobility Predictor (AMPPRO) score: 27-42 collected within the last 24 months
* Ability to read, write, and understand English.

Exclusion Criteria:

* Any health condition that would prevent safely completing trial activities.
* Any individuals that weigh 275 lbs or more.
* Any individuals who wear their prosthesis less than 3 days a week or less than a total of 24 hours a week
* Individuals with a history of acute or chronic residual limb breakdown
* Individuals with declining health status such that he/she subsequently reports reduced activity over the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-11 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Prosthetic Limb Users Survey of Fall-Related Self-Efficacy (PLUS-F-SEF) | Collected at baseline, 1-month, 3-month, 6-month, 9-month, and 12-month assessments.
  The PLUS-F-SEF is a 15-item self-report instrument we developed in the present study to measure perceived ability to avoid a loss of balance while performing an activity. Respondents rate their degree of confidence on a 5-point scale from "not at all confident" (1) to "very much confident" (5). A standardized T-score is generated for the PLUS-F-SEF using a lookup table that converts the raw score to a T-score.
Prosthetic Limb Users Survey of Fall-Related Anxiety (PLUS-F-ANX) | Collected at baseline, 1-month, 3-month, 6-month, 9-month, and 12-month assessments.
  The PLUS-F-ANX is a 15-item self-report instrument we developed in the present study to measure perceived apprehensions or concerns about losing one's balance or falling. Respondents rate the frequency with which they experience various emotional responses on a 5-point scale from "never" (1) to "always" (5). A standardized T-score is generated for the PLUS-F-ANX using a lookup table that converts the raw score to a T-score.
Prosthetic Limb Users Survey of Fall-Related Avoidance Behaviors (PLUS-F-AVB) | Collected at baseline, 1-month, 3-month, 6-month, 9-month, and 12-month assessments.
  The PLUS-F-AVB is a 15-item self-report instrument we developed in the present study to measure perceived changes in the manner or frequency with which activities are performed to avoid losing one's balance or falling. Respondents rate the frequency with which they make changes on a 5-point scale from "never" (1) to "always" (5). A standardized T-score is generated for the PLUS-F-AVB using a lookup table that converts the raw score to a T-score.
Prosthetic Limb Users Survey of Fall-Related Interference (PLUS-F-INT) | Collected at baseline, 1-month, 3-month, 6-month, 9-month, and 12-month assessments.
  The PLUS-F-INT is a 15-item self-report instrument we developed in the present study to measure perceived restrictions in social, cognitive, emotional, and/or physical life situations due to risk of falls. Respondents rate the amount of interference on a 5-point scale from "not at all" (1) to "very much" (5). A standardized T-score is generated for the PLUS-F-INT using a lookup table that converts the raw score to a T-score.
Number of Reported Falls and Near-Fall Events | Collected every two weeks starting at baseline up to 12 months
  Participants will be contacted every 2 weeks starting at baseline through study completion to determine whether they experienced a fall event (either a fall or near-fall). For each event experienced, participants will be asked to report the details of that event using the Lower Limb Prosthesis User Fall Event Survey we developed in a prior study. This instrument asks respondents to report the activity, surroundings, situation, mechanics, and consequences of each event. Fall events will be scored as the total number of falls, near-falls, and all fall events experienced. The details of the events are descriptive in nature and will be used to characterize the falls experienced by the participant.

SECONDARY OUTCOMES:
EuroQol 5 Dimensions (EQ-5D) | Collected at baseline, 6-month, and 12-month assessments.
  The EQ-5D is a self-report measure of health-related quality of life (HRQL). The EQ-5D includes a descriptive component and a visual analog scale (VAS). The descriptive component evaluates respondents' HRQL in five areas (i.e., mobility, self-care, usual activities, pain/discomfort, and anxiety/depression) using a five- or three-level response option. We will use the five-level response option (EQ-5D-5L) for this study, where level 1 indicates "no problem" and level 5 indicates "unable to/extreme problems." The VAS component measures the respondent's HRQL on a 0 (the worst imaginable health) to 100 (the best imaginable health) VAS scale.
Balance Recovery Scale (BRC) | Collected at baseline, 6-month, and 12-month assessments.
  The BRC is a 19-item self-report questionnaire designed to measure balance recovery self-efficacy (i.e., perceived reactive balance recovery). Respondents rate the degree of confidence with which they can recover from different losses of balance on a 10-point scale, from "cannot do at all" (0) to "highly certain can do" (10). A summary score is generated from the responses to questions in the BRC.
Fear of Falling Avoidance Behaviors Questionnaire (FFABQ) | Collected at baseline, 6-month, and 12-month assessments.
  The FFABQ is a 14-item self-report instrument that measures the degree to which respondents avoid activities due to their fear of falling. Respondents rate the amount of times they avoid select activities due to their fear of falling on a 5-point scale from "always (100% of the time)" to "never (0% of the time)." A summary score is generated from the responses to questions in the FFABQ.
Prosthetic Limb Users Survey of Mobility (PLUS-M) | Collected at baseline, 6-month, and 12-month assessments.
  The PLUS-M is a 12-item self-report instrument we developed in a prior study to measure mobility with an LLP. Respondents rate their perceived difficulty with performing various household and community activities on a 5-point scale, ranging from "without any difficulty" (5) to "unable to do" (1). A standardized T-score is generated for the PLUS-M using a lookup table that converts the raw score to a T-score.
Timed Up and Go (TUG) | Collected at baseline, 6-month, and 12-month assessments.
  The TUG is a performance-based test designed to measure basic mobility tasks, such as sit-to-stand, gait initiation, walking, turning, and stand-to-sit. The TUG requires the participant stand up from a standard chair with arms, walk at a comfortable speed for 3 meters, turn around, and return to sit in the chair. The administrator times the participant as they perform the test. Lower TUG times are indicative of better performance (mobility). The TUG is scored as the lowest time achieved in one of two timed trials.
Ten Meter Walk Test (10mWT) | Collected at baseline, 6-month, and 12-month assessments.
  The 10mWT is a performance-based test designed to measure a participant's self-selected walking speed. The 10mWT requires the participant to walk at a normal speed between lines taped on the floor. The administrator measures the time required to walk the middle six meters of the 10-meter distance. Lower times (ie, faster speed) is indicative of better performance. The 10mWT is scored by calculating the participant's walking speed in meters per second (m/s).
Two Minute Walk Test (2MWT) | Collected at baseline, 6-month, and 12-month assessments.
  The 2MWT is a performance test designed to measure submaximal walking endurance. The 2MWT requires the participant to walk as far as possible over a period of 2 minutes. Longer distances indicate better performance (i.e., greater endurance). The administrator measures the distance the participant travels during the test. The 2MWT is scored as the total distance traveled in meters (m) over the test period.

CONTACTS AND LOCATIONS:
Overall Officials: Shane R. Wurdeman, PhD, Principal Investigator — Hanger Institute for Clinical Research and Education
Locations (1):
- Hanger Inc., Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hu LY, Huang MW, Ke SW, Tsai CF. The distance function effect on k-nearest neighbor classification for medical datasets. Springerplus. 2016 Aug 9;5(1):1304. doi: 10.1186/s40064-016-2941-7. eCollection 2016. PMID 27547678
- [Background] Berry D. Microprocessor prosthetic knees. Phys Med Rehabil Clin N Am. 2006 Feb;17(1):91-113, vii. doi: 10.1016/j.pmr.2005.10.006. PMID 16517347
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Efird J. Blocked randomization with randomly selected block sizes. Int J Environ Res Public Health. 2011 Jan;8(1):15-20. doi: 10.3390/ijerph8010015. Epub 2010 Dec 23. PMID 21318011
- [Background] Eberly VJ, Mulroy SJ, Gronley JK, Perry J, Yule WJ, Burnfield JM. Impact of a stance phase microprocessor-controlled knee prosthesis on level walking in lower functioning individuals with a transfemoral amputation. Prosthet Orthot Int. 2014 Dec;38(6):447-55. doi: 10.1177/0309364613506912. Epub 2013 Oct 17. PMID 24135259
- [Background] Hafner BJ, Smith DG. Differences in function and safety between Medicare Functional Classification Level-2 and -3 transfemoral amputees and influence of prosthetic knee joint control. J Rehabil Res Dev. 2009;46(3):417-33. PMID 19675993
- [Background] Hafner BJ, Willingham LL, Buell NC, Allyn KJ, Smith DG. Evaluation of function, performance, and preference as transfemoral amputees transition from mechanical to microprocessor control of the prosthetic knee. Arch Phys Med Rehabil. 2007 Feb;88(2):207-17. doi: 10.1016/j.apmr.2006.10.030. PMID 17270519
- [Background] Jepson F, Datta D, Harris I, Heller B, Howitt J, McLean J. A comparative evaluation of the Adaptive knee and Catech knee joints: a preliminary study. Prosthet Orthot Int. 2008 Mar;32(1):84-92. doi: 10.1080/03093640701676376. PMID 18330807
- [Background] Kahle JT, Highsmith MJ, Hubbard SL. Comparison of nonmicroprocessor knee mechanism versus C-Leg on Prosthesis Evaluation Questionnaire, stumbles, falls, walking tests, stair descent, and knee preference. J Rehabil Res Dev. 2008;45(1):1-14. doi: 10.1682/jrrd.2007.04.0054. PMID 18566922
- [Background] Pauley T, Devlin M, Heslin K. Falls sustained during inpatient rehabilitation after lower limb amputation: prevalence and predictors. Am J Phys Med Rehabil. 2006 Jun;85(6):521-32; quiz, 533-5. doi: 10.1097/01.phm.0000219119.58965.8c. PMID 16715022
- [Background] Wong CK, Chihuri ST, Li G. Risk of fall-related injury in people with lower limb amputations: A prospective cohort study. J Rehabil Med. 2016 Jan;48(1):80-5. doi: 10.2340/16501977-2042. PMID 26694526
- [Background] Pezzin LE, Dillingham TR, MacKenzie EJ. Rehabilitation and the long-term outcomes of persons with trauma-related amputations. Arch Phys Med Rehabil. 2000 Mar;81(3):292-300. doi: 10.1016/s0003-9993(00)90074-1. PMID 10724073
- [Background] McWhinnie DL, Gordon AC, Collin J, Gray DW, Morrison JD. Rehabilitation outcome 5 years after 100 lower-limb amputations. Br J Surg. 1994 Nov;81(11):1596-9. doi: 10.1002/bjs.1800811110. PMID 7827880
- [Background] van Velzen JM, van Bennekom CA, Polomski W, Slootman JR, van der Woude LH, Houdijk H. Physical capacity and walking ability after lower limb amputation: a systematic review. Clin Rehabil. 2006 Nov;20(11):999-1016. doi: 10.1177/0269215506070700. PMID 17065543
- [Background] Wong CK, Rheinstein J, Stern MA. Benefits for Adults with Transfemoral Amputations and Peripheral Artery Disease Using Microprocessor Compared with Nonmicroprocessor Prosthetic Knees. Am J Phys Med Rehabil. 2015 Oct;94(10):804-10. doi: 10.1097/PHM.0000000000000265. PMID 25768067
- [Background] Kim J, Major MJ, Hafner B, Sawers A. Frequency and Circumstances of Falls Reported by Ambulatory Unilateral Lower Limb Prosthesis Users: A Secondary Analysis. PM R. 2019 Apr;11(4):344-353. doi: 10.1016/j.pmrj.2018.08.385. Epub 2019 Jan 15. PMID 30195705
- [Background] Miller WC, Speechley M, Deathe B. The prevalence and risk factors of falling and fear of falling among lower extremity amputees. Arch Phys Med Rehabil. 2001 Aug;82(8):1031-7. doi: 10.1053/apmr.2001.24295. PMID 11494181
- [Background] Gauthier-Gagnon C, Grise MC, Potvin D. Enabling factors related to prosthetic use by people with transtibial and transfemoral amputation. Arch Phys Med Rehabil. 1999 Jun;80(6):706-13. doi: 10.1016/s0003-9993(99)90177-6. PMID 10378500
- [Background] Legro MW, Reiber G, del Aguila M, Ajax MJ, Boone DA, Larsen JA, Smith DG, Sangeorzan B. Issues of importance reported by persons with lower limb amputations and prostheses. J Rehabil Res Dev. 1999 Jul;36(3):155-63. PMID 10659798
- [Background] Highsmith MJ, Kahle JT, Bongiorni DR, Sutton BS, Groer S, Kaufman KR. Safety, energy efficiency, and cost efficacy of the C-Leg for transfemoral amputees: A review of the literature. Prosthet Orthot Int. 2010 Dec;34(4):362-77. doi: 10.3109/03093646.2010.520054. Epub 2010 Oct 24. PMID 20969495
- [Background] Sawers AB, Hafner BJ. Outcomes associated with the use of microprocessor-controlled prosthetic knees among individuals with unilateral transfemoral limb loss: a systematic review. J Rehabil Res Dev. 2013;50(3):273-314. doi: 10.1682/jrrd.2011.10.0187. PMID 23881757
- [Background] Kaufman KR, Bernhardt KA, Symms K. Functional assessment and satisfaction of transfemoral amputees with low mobility (FASTK2): A clinical trial of microprocessor-controlled vs. non-microprocessor-controlled knees. Clin Biomech (Bristol). 2018 Oct;58:116-122. doi: 10.1016/j.clinbiomech.2018.07.012. Epub 2018 Jul 19. PMID 30077128
- [Background] Stevens PM, Wurdeman SR. Prosthetic Knee Selection for Individuals with Unilateral Transfemoral Amputation: A Clinical Practice Guideline. J Prosthet Orthot. 2019 Jan;31(1):2-8. doi: 10.1097/JPO.0000000000000214. Epub 2018 Nov 9. PMID 30662248
- [Background] Kannenberg A, Zacharias B, Probsting E. Benefits of microprocessor-controlled prosthetic knees to limited community ambulators: systematic review. J Rehabil Res Dev. 2014;51(10):1469-96. doi: 10.1682/JRRD.2014.05.0118. PMID 25856664
- See also: (CMS), U. S. C. f. M. m. S. Lower limb prosthetic workgroup consensus document (September 2017). — https://www.cms.gov/Medicare/Coverage/DeterminationProcess/downloads/LLP_Consensus_Document.pdf